CLINICAL TRIAL: NCT05147103
Title: Investigation of the Duration of Low-intensity Focused Ultrasound
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-892
Record Dates: First submitted 2021-11-10; First posted 2021-12-07 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Development of LIFU for Clinical Purposes
Keywords: low-intensity focused ultrasound; transcranial magnetic stimulation

STUDY DESIGN:
Intervention Model Description: Multi-visit study, testing various LIFU durations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Duration Trials (Experimental): Six different durations (three intermittent and three continuous) of LIFU application will be tested across six study sessions. Response recorded using TMS and EMG.
  Interventions: Device: Low-Intensity Focused Ultrasound

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound — LIFU application using various durations, responses of neuromodulation recorded using TMS and EMG.

SUMMARY:
This project examines the effects of various durations of noninvasive neuromodulation on muscle contractions. The investigators believe this study will help to better understand noninvasive brain stimulation techniques that may have the potential to aid in addiction, pain, and mental health issues. Participants undergo structural imaging, a functional Magnetic Resonance Image (fMRI) and computed tomography (CT). These images are used to align the low-intensity focused ultrasound (LIFU) and transcranial magnetic stimulation (TMS) devices to temporarily change brain activity. Electromyography (EMG) will be used to record muscle contractions of the hand.

ELIGIBILITY:
Inclusion Criteria:

* Above criteria and must understand and speak English.

Exclusion Criteria:

* Contraindications to MRI, CT, or TMS

  1. Claustrophobia
  2. Pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
  3. Pregnancy
  4. Active medical disorder or treatment with potential CNS effects
  5. History of neurologic disorder
  6. History of head injury resulting in loss of consciousness for >10 minutes
  7. History of alcohol or drug dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Waveforms | Outcomes assessed throughout participation - an average of 3 weeks.
  Changes in waveform peak will be observed per each variable application of LIFU

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legon W, Bansal P, Tyshynsky R, Ai L, Mueller JK. Transcranial focused ultrasound neuromodulation of the human primary motor cortex. Sci Rep. 2018 Jul 3;8(1):10007. doi: 10.1038/s41598-018-28320-1. PMID 29968768
- [Background] Legon W, Ai L, Bansal P, Mueller JK. Neuromodulation with single-element transcranial focused ultrasound in human thalamus. Hum Brain Mapp. 2018 May;39(5):1995-2006. doi: 10.1002/hbm.23981. Epub 2018 Jan 29. PMID 29380485
- [Background] Legon W, Sato TF, Opitz A, Mueller J, Barbour A, Williams A, Tyler WJ. Transcranial focused ultrasound modulates the activity of primary somatosensory cortex in humans. Nat Neurosci. 2014 Feb;17(2):322-9. doi: 10.1038/nn.3620. Epub 2014 Jan 12. PMID 24413698